CLINICAL TRIAL: NCT05992376
Title: Impact Evaluation of the Global Alliance for Improved Nutrition (GAIN) Vegetables for All Program in Kenya
Brief Title: Vegetables for All Evaluation Kenya
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Kula Vyema Centre of Food Economics (Unknown); Jomo Kenyatta University of Agriculture and Technology (JKUAT) (Unknown)
Responsible Party: Principal Investigator, Valerie Flax, Senior Research Public Health Analyst, RTI International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 424604
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Vegetable Consumption
Keywords: diet; vegetables; market intervention; social and behavior change communication intervention; children; Kenya

STUDY DESIGN:
Intervention Model Description: Data will be collected through household surveys, mama mboga surveys, in-depth interviews (IDIs), and focus group discussions (FGDs). The protocol team has selected a subset of intervention FFZs for the evaluation and identified an equal number of geographic areas of similar size and level of urbanicity to serve as the controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Food system and demand generation
- Control/No Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Food system and demand generation — The Vegetables for All program will create FitFood Zones (FFZs) in low-income estates in urban and peri-urban areas with a minimum of 1,000 households and 10 mama mbogas. FFZs are the last mile/point of purchase for delivering a variety of fresh, safe, and accessible vegetables to BoP households. The program will support mama mbogas to source vegetables from Good Agricultural Practices (GAP)-compliant suppliers, support the uptake of digital solutions for mama mbogas to access vegetables, create business-to-business mentorship opportunities, and support county governments to improve market infrastructure. To encourage BoP parents of children 3-11 years to buy and consume more vegetables, the program will include a demand generation component. This will be implemented through a communication campaign, including above-the-line (ATL) activities (mass media such as radio and television), below-the-line (BTL) activities (market activations and others), and FFZ branding.
  Arms: Intervention

SUMMARY:
Global Alliance for Improved Nutrition (GAIN)'s "Vegetables for All" program in Kenya seeks to improve consumption of healthy foods by improving supply, increasing demand, and improving the enabling environment for different vegetables by operating at multiple levels - individuals, households, markets, producers, and policies. RTI and local partners propose to conduct impact and process evaluations of GAIN's program tailored to the theory of change. The evaluation will include a mix of quantitative and qualitative methods and will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) evaluation framework.

DETAILED DESCRIPTION:
Background: In urban and peri-urban areas in Kenya, Consumption of vegetables is low in bottom of pyramid (BoP) households, which earn < 3.20 US dollars per person per day. To increase vegetable consumption in this population, GAIN will implement the Vegetables for All program, which aims to improve access to safe and fresh vegetables in Fit Food Zones (FFZs) and to generate demand for vegetables through a radio/television campaign and FFZ branding. The main retailers in the FFZ are mama mbogas (vegetable vendors), who will be linked to suppliers that are Good Agricultural Practices (GAP) compliant.

Objective: The overall objectives of the evaluation are: 1) to assess the effectiveness of GAIN's Vegetables for All program for increasing the quantity of vegetables consumed and improving the diet quality of BoP consumers and 2) to conduct a process evaluation of GAIN's program that provides data to support findings of the impact evaluation.

Methods: This study will use a mixed-methods quasi-experimental design in which 124 FFZs are assigned to intervention or control in Nairobi, Kiambu, Machakos, Mombasa, and Nakuru counties. The impacts will be assessed through cross-sectional population-based surveys of households with women 18-49 years who have a child 3-11 years in 62 intervention and 62 control FFZs at baseline and endline (N=1,364 at each time point). Mama mboga surveys will be conducted in all 124 sampled FFZs at baseline, midline, and endline (N=372 at each time point). Qualitative data will be collected at midline and endline. In-depth interviews (IDIs) will be conducted with vegetable value chain actors and other stakeholders (N=18 at each time point). Focus group discussions (FGDs) will be conducted with mama mbogas (20 FGDs at each time point) and household members (20 FGDs at each time point). The analysis will be performed using difference-in-difference estimation (surveys) and thematic content analysis methods (qualitative).

ELIGIBILITY:
Household Surveys

Inclusion Criteria:

* Reside in the FFZs assigned;
* Be a woman between 18-49 years old;
* Have a child 3-12 years old
* The household earns <$3.20 per person per day;
* Be able to speak one of the main local languages and/or Kiswahili;
* Provide informed consent to participate in the study.

Mama Mboga Surveys

Inclusion Criteria:

* Be a mama mboga retailer of vegetables in a FFZ in the districts selected for the evaluation;
* Be in business for at least 6 months
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Kiswahili;
* Provide informed consent to participate in the study.

In-depth interviews with value chain actors

Inclusion criteria:

* Be a vegetable supplier to mama mbogas as part of the FFZ, are involved in demand generation activities, or involved in food safety compliance;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Kiswahili;
* Provide informed consent to participate in the study.

Focus group discussion (FGD) participants will be selected from lists of participants in the FFZ and household surveys and will be consented again for the FGDs if they meet the following criteria:

FGDs with households

Inclusion criteria:

* Be a woman living in a BoP household in a FFZ selected for the evaluation;
* Have ever visited a mama mboga's place of business
* Participated in the baseline survey
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Kiswahili;
* Provide informed consent to participate in the study.

FGDs with mama mbogas

Inclusion criteria:

* Be a mama mboga linked to the Vegetables for All project in one of the intervention FFZs
* Have been a mama mboga for at least 6 months
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Kiswahili;
* Provide informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4680 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Grams of Vegetables Consumed | Baseline (September 2023), endline (September 2025) (2 years)
  Change in the mean grams of vegetables consumed during the last 24 hours by children 3-11 years old in BoP households in Fit Food Zones

CONTACTS AND LOCATIONS:
Overall Officials: Simon Kimenju, PhD, MSc, Principal Investigator — Kula Vyema Centre of Food Economics
Locations (1):
- Kula Vyema Centre of Food Economics, Kiambu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be shared through Nesstar.